CLINICAL TRIAL: NCT02074787
Title: A Comparison of Three Non-invasive Imaging Modalities (Thermography, Laser Doppler and SIAscope) for the Assessment of Adult Burns Injuries
Brief Title: Imaging of Adult Burn Injuries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Royal College of Surgeons of England (Unknown)
Responsible Party: Sponsor
Other Study IDs: C&W13/090; 14/EE/0048 (Other: Regional Ethics Committee (UK)); 141406 (Other: IRAS project ID)
Record Dates: First submitted 2014-02-27; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Thermography; Laser Doppler Blood Flow; Spectrophotometric Intracutaneous Analysis
MeSH Terms: interventions — Thermography; Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult burn injuries: Adult patients with burns injuries attending the regional burns unit at Chelsea & Westminster hospital between 48 and 72 hours post burn will be invited to take part in the study at the time of presentation to the unit.
  Interventions: Device: Thermography; Device: Laser Doppler; Device: Spectrophotometric Intracutaneous analysis

INTERVENTIONS:
Device: Thermography — Standard thermographic images
  Other Names: FLIR E50mx
Device: Laser Doppler — standard laser doppler analysis
  Other Names: Moor systems laser doppler blood flow analysis
Device: Spectrophotometric Intracutaneous analysis — standard SIA scope imaging
  Other Names: SIA scope

SUMMARY:
Burn injuries are a common presentation to A&E in the UK (175,000 per year) of whom 13,000 require hospital admission. Treatment of a single burn can cost more than £63,000, and is ultimately dependent on the depth. Most burns are assessed by experienced clinicians within a few days of injury. Accurate evaluation of burn depth can be very difficult with the naked eye. Inaccuracy can lead to longer hospital stays, worse scarring and greater financial costs for the NHS. Where the burn depth (and the degree of damage to the underlying blood supply of the skin) is not clear by visual inspection, adjuncts may be used to aid clinical decision-making. Currently, the "gold standard" method of assessing skin blood flow in order to help burn specialists in their assessment of burn depth is Laser Doppler Imaging (LDI). However, LDI machines can be very large, slow to collect the images, and a single imaging unit costs roughly £50,000. Consequently their use is restricted to the assessment of small burns in compliant patients treated in specialist units. Thermal imaging (thermography) has evolved rapidly as a useful diagnostic tool in many medical disciplines. Previous studies have shown that there are significant changes in skin physiology (such as temperature and pigmentation) depending on the depth of the burn. Portable, high-resolution thermal cameras are now affordable, easy to use and can provide numerical results in under a second. Similarly, measurement of skin pigment levels can be achieved using portable devices such as the Spectrophotometric Intracutaneous analysis scope (SIAscope). The aim of this study is to determine if alternative measures such as thermography or SIAscope can be as useful in the assessment of adult burns as LDI currently is. If this study demonstrates this then these results will inform further studies that would investigate these alternative imaging methods as a diagnostic and prognostic tool in the management of burns not only in adults but also in children presenting to non-specialised units such as A&E.

DETAILED DESCRIPTION:
Adult acute burn injuries are currently "read" by experienced clinicians at 2-3 days post injury in order to determine the necessary treatment and likely clinical outcome. Adjuncts to this process aim to inform the clinician of structural damage to the sub dermal vasculature. The current gold standard investigation is laser doppler imaging (LDI) of dermal blood flow. However, due to time and resource constraints, this technique is often only applied to dermal burns of indeterminate thickness. Thermography and the SIAscope potential offer quicker, quantitative analysis with equipment currently in routine medical use in other clinical disciplines.

To validate its use against the current gold standard (LDI)burns of variable thicknesses will need to be assessed and compared with clinical outcome. Consequently, in this study, patients with superficial burns that would not usually require LDI will be included for comparison. All patients will be reassured that thermography, the SIAscope and LDI are non-invasive, non-harmful, quick and will not affect their burn management in any way. Images will be labelled by an anonymised study number and stored in on secure hospital servers according to the Trust's information governance policy.

ELIGIBILITY:
Inclusion Criteria:

* adults burn injury within 72 hours of presentation able to undergo all three imaging modalities

Exclusion Criteria:

* children patients not consenting

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with burns injuries attending the regional burns unit at Chelsea & Westminster hospital between 48 and 72 hours post burn will be invited to take part in the study at the time of presentation to the unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
95% healing | within 4 weeks of presentation
  The time to 95% epithelial healing of adult burn injuries as assessed by experienced burns clinicians

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea & Westminster NHS Foundation Trust, London, London, United Kingdom